CLINICAL TRIAL: NCT00338390
Title: Study of Changes in CD4 Lymphocyte Count in Patients With a HAART Regimen Including DDI + Tenofovir and With Viral Suppression Following the Replacement of Tenofovir With Abacavir Once Daily or Following the Double Replacement of DDI + Tenofovir With Abacavir + Lamivudine in a Single Tablet
Brief Title: Study to Evaluate Changes in CD4 on Replacing TDF With ABC or DDI+TDF With ABC+3TC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUROPA; 2004-003749-42
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infections
Keywords: Antiretrovirals; CD4 cell count; toxicity
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Didanosine; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Maintain antiretroviral treatment
- 2 (Experimental): Change tenofovir to abacavir and increase didanosine dose to 400 mg/day if weight is > 60 Kg. or to 250mg/day if weight is < 60 kg.
  Interventions: Drug: Abacavir; Drug: Didanosine
- 3 (Experimental): Change tenofovir and didanosine to abacavir + lamivudine (600mg+300 mg/day in one single tablet).
  Interventions: Drug: Abacavir+Lamivudine

INTERVENTIONS:
Drug: Abacavir — Change tenofovir to abacavir
  Other Names: n/h.
  Arms: 2
Drug: Didanosine — Increase didanosine dose to 400 mg/day if weight is > 60 Kg. or to 250mg/day if weight is < 60 kg.
  Other Names: n/h.
  Arms: 2
Drug: Abacavir+Lamivudine — Change tenofovir and didanosine to abacavir + lamivudine (600mg+300 mg/day in one single tablet).
  Other Names: n/h.
  Arms: 3

SUMMARY:
The study aims to ascertain whether the sole replacement of tenofovir with abacavir once a day improves the immunological response obtained with tenofovir + ddI or whether it is better to perform a double replacement of tenofovir and ddI with abacavir + lamivudine (joint formulation) in a single daily dose to achieve these objectives.

DETAILED DESCRIPTION:
Different works have shown a high rate of virological failure among patients on abacavir + lamivudine + tenofovir or ddI + 3TC + tenofovir, thus rendering the use of these combinations actively unadvisable.

Furthermore, recent studies have also shown that ABC+3TC are associated with a significantly higher increase in CD4 than the current treatment standard formed by AZT+3TC. This provides us with grounds to suppose that patients with TDF+ddI may recover their CD4 with ABC+3HT. Similarly, and recently, the existence of pharmacokinetic interactions between tenofovir + abacavir has begun to be questioned.

Finally, the replacement of tenofovir with abacavir or tenofovir + ddI with abacavir + lamivudine does not detract from the potency of HAART, the toxicity profile is different and their behaviour at mitochondrial level is similar.

This study aims to ascertain whether the sole replacement of tenofovir with abacavir once a day improves the immunological response obtained with tenofovir + ddI or whether it is better to perform a double replacement of tenofovir and ddI with abacavir + lamivudine (joint formulation) in a single daily dose to achieve these objectives.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* HIV-1 infected patients.
* Patients on triple HAART therapy including ddI + tenofovir plus a PI or NNRTI for at least 3 months.
* Patients with an undetectable HIV-1 viral load (< 50 copies RNA / mL or < centre's limit of detection) over the last 6 months.
* Not be on treatment with immunosuppressives, such as: hydroxyurea, interferon, ribavirin or cytostatics.
* Not be on treatment with interleukin-2 or other immunomodulators.
* Women may not be of fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or must undertake to use a barrier contraceptive method during the study.
* Signature of the informed consent.

Exclusion Criteria:

* Incapacity to give informed consent.
* Bad adherence or treatment interruptions over the previous 6 months.
* Prior exposure to abacavir.
* HAART Therapy including ddI at a dose of 400mg + tenofovir if weight > 60 kg or ddI 250 mg + tenofovir if weight < 60 kg.
* Suspicion of cross resistances to abacavir and lamivudine.
* Hepatic or pancreatic analytical alterations 4 times above the limit of normality.
* Presence of opportunistic infections and/or recent tumours (< 6 months).
* Patients participating in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that increase their number of CD4 lymphocytes with regard to the baseline. | At 12, 24, 36 and 48 weeks

SECONDARY OUTCOMES:
To evaluate the proportion of patients with viral load of HIV-1 <50 copies of the combinations studied during the follow-up period. | At 12, 24, 36 and 48 weeks.
Incidence of new clinical adverse events that appear . | during 48 weeks of follow-up
Evolution of the clinical adverse events that were already present at the time they were included in the study. | during the 48 weeks of follow-up
Rate of treatment drop-outs due to the appearance of adverse events | during the 48 weeks of follow-up
Incidence of new laboratory alterations that appear during the follow-up period (change in renal parameters, changes in lactate levels, modification of pancreatic enzymes, changes in lipid parameters). | during the follow-up period
Evolution of the laboratory alterations that were already present at the time they were included in the study. | during the 48 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Enric Pedrol, MD, PhD, Principal Investigator — Fundació Hospital de Granollers
Locations (21):
- Spain (21):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Sant Jaume de Calella, Calella, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Basurto, Bilbao, Bilabao
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Sierrallana, Torrelavega, Cantabria
  - Hospital General de Castellón, , Castellón,, Castelló, Castello
  - H. del S.A.S. Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - H. San Fco Borja Gandia, Gandia, Gandia
  - Hospital de Cabueñes, Gijón, Gijon
  - Hospital Clínico San Cecílio, Granada, Granada
  - Fundació Hospital de Granollers,, Barcelona, Granollers
  - Hospital Arquitecto Marcide, Ferrol, La Coruña
  - Fundación Jiménez Diaz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Virgen Macarena, Seville, Sevilla
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Xeral de Vigo, Vigo, Vigo